CLINICAL TRIAL: NCT02055209
Title: Genomics, Environmental Factors and Social Determinants of Cardiovascular Disease in African-Americans Study (GENE-FORECAST)
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 140048; 14-HG-0048
Record Dates: First submitted 2014-02-04; First posted 2014-02-05 (Estimated); Last update posted 2026-02-05 (Actual); Status verified 2025-11-18

CONDITIONS: Hypertension
Keywords: African American; Natural History
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: Adults only, all genders, US born African American

SUMMARY:
Our objective is to develop a community-based cohort and novel genomic science resource for defining the biological significance of ancestry-related genomic variation in African-Americans within the GENE-FORECAST :GENomics, Environmental FactORs and the Social DEterminants of Cardiovascular Disease in African Americans STudy. AIM I. examine the associations between common or ancestry-related DNA variants and CVD risk factors (e.g. hypertension) and phenotypes (e.g. coronary artery calcification) in African-Americans (AA).AIM II. To examine the associations between health behaviors or social-environmental factors and CVD risk factors and phenotypes in AA.The study is designed to create a cohort amenable to nested case-control analyses based on a community-based sampling frame with a target size of approximately 1800 self-identified, US -born, African-American (AA) men and women (ages 21-65) to be recruited over the next 5-6 years from the metropolitan Washington DC, Montgomery County (MC) and Prince George s County (PG) areas to be recruited to the NIH Clinical Center. The initial participant recruitment two approaches: 1) a random-digit telephone screening survey targeting study-eligible AA that will be consented and invited to an evaluation visit in the NIH Clinical Center which we contracted with a well-established survey group (Southern Research Group [SRG]); and 2) a community outreach effort to recruit participants into the Clinical Center by leveraging marketing and the engagement of community-based leaders, organizations and faith-based institutions in the area. this approach will yield a sample with normal individuals as well as a high proportion of AA with CVD risk factors such as obesity and hypertension that predispose to the eventual clinical signs and symptoms of CVD (e.g. heart attack and stroke). it is anticipated that the prevalence of clinically manifest CVD (history of angina, heart attack or stroke) will be less than 10-15% of the sample. All will medical evaluation (e.g. anthropometrics, blood pressure), laboratory tests (e.g. lipid levels, kidney function), social determinants profiles (e.g. socioeconomic status (SES), perceived stress, discrimination, depression, perceived neighborhood characteristics), blood/urine collection for deep-sequencing based omic analyses (e.g. whole exome sequencing, and RNA-Seq), as well as testing for pre-clinical , biomarkers of the pathobiological processes of CVD or CVD phenotypes (e.g. coronary artery calcification, microalbuminuria, leukocyte telomeres, or vascular dysfunction). It is anticipated that these deep sequencing efforts will yield novel ancestry-related DNA variants associated with the CVD phenotypes; yet with unclear biological significance in elucidating racial disparities in CVD. Accordingly, our protocol also includes a Genotype-to-Phenotype (G2P) component that re- contacts subsets of the cohort based on their genotype (e.g. APOL1 chronic kidney disease risk alleles) for a call-back visit for more in-depth phenotyping and characterization of the potential effect of the DNA variant of interest on human systems biology. In some cases family members of the proband may also be invited to participate in these G2P studies to further characterize the biological significance of these putative functional DNA variants of interest.

The primary outcome variables involve well established CVD phenotypes: 1) CVD risk factors (e.g. hypertension, dyslipidemia), 2) markers of pre-clinical CVD (i.e. coronary artery calcification, coronary plaque burden by cardiac CT angiography (CTA), carotid plaque burden by 3D ultrasound, vascular dysfunction, microalbuminuria, C-reactive protein, Vitamin D levels). The protocol will assess exposures associated with CVD and relevant covariates including: 1) social determinants (e.g. socioeconomic status (SES), perceived stress, discrimination, and depression); 2) environmental factors such as neighborhood characteristics (geospatial features of healthy lifestyles [e.g. walkability]) and 3) behavioral factors (e.g. diet, physical activity). The G2P callback visit protocol will involve additional measures of in-depth phenotyping that include: 1) peripheral immune cell phenotyping (e.g. T-cell, monocyte subsets); 2) blood/immune cell RNAseq; 3) iPSC cell line generation (endothelial; vascular smooth muscle cells) and analysis of cardiovascular cell systems biology; 4) HDL proteome analysis, 5) FDG PET/CT and/or PET/MRI scan (vascular inflammation) 6) echocardiography, 7) bisulfite sequencing for identifying sites of DNA methylation, and 8) chromatin immunoprecipitation followed by sequencing (Chip-Seq) for identifying sites of histone modification. It is anticipated that this multi-level, multi-dimensional analysis of genomic and phenotypic characteristics of AA will advance our understanding of the bio-social determinants of the intragroup variance and the increased overall burde...

DETAILED DESCRIPTION:
Our objective is to develop a community-based cohort and novel genomic science resource for defining the biological significance of ancestry-related genomic variation in African-Americans within the GENE-FORECAST :GENomics, Environmental FactORs and the Social DEterminants of Cardiovascular Disease in African Americans STudy. This resource will enable our team to test the working hypothesis that race-ancestry differences in the burden of cardiovascular disease (CVD) reflects the influence of a unique interplay between the distinct genomic variation characteristic of African-Americans (AA) and the exposome of social determinants and environmental factors that influence the pathogenesis of CVD in AA. The specific aims are:

AIM I. To examine the associations between common or ancestry-related DNA variants and CVD risk factors (e.g. hypertension) and phenotypes (e.g. coronary artery calcification) in African-Americans (AA).

AIM II. To examine the associations between health behaviors or social-environmental factors and CVD risk factors and phenotypes in AA.

The study is designed to create a cohort amenable to nested case-control analyses based on a community-based sampling frame with a target size of approximately 1800 self-identified, US -born, African-American (AA) men and women (ages 21-65) to be recruited over the next 5-6 years from the metropolitan Washington DC, Montgomery County (MC) and Prince George s County (PG) areas to be recruited to the NIH Clinical Center. The initial participant recruitment strategy involved two approaches: 1) a random-digit telephone screening survey targeting study-eligible AA that will be consented and invited to an evaluation visit in the NIH Clinical Center which we contracted with a well-established survey group (Southern Research Group [SRG]); and 2) a community outreach effort to recruit participants into the Clinical Center by leveraging marketing and the engagement of community-based leaders, organizations and faith-based institutions in the area. We are no longer contracting with SRG but rather focusing on community outreach and marketing for recruitment to the Clinical Center. The contract with SRG was terminated after the first two years of the protocol due to low yield of recruitment to the Clinical Center compared to community outreach.

Given the high burden of CVD among AA, this approach will yield a sample with normal individuals as well as a high proportion of AA with CVD risk factors such as obesity and hypertension that predispose to the eventual clinical signs and symptoms of CVD (e.g. heart attack and stroke). Based on previous epidemiology studies, this protocol s participant ascertainment approach and the target demographic profile; it is anticipated that the prevalence of clinically manifest CVD (history of angina, heart attack or stroke) will be less than 10-15% of the sample. All participants will undergo extensive evaluation in the Clinical Center that includes: medical evaluation (e.g. anthropometrics, blood pressure), laboratory tests (e.g. lipid levels, kidney function), social determinants profiles (e.g. socioeconomic status (SES), perceived stress, discrimination, depression, perceived neighborhood characteristics), blood/urine collection for deep-sequencing based omic analyses (e.g. whole exome sequencing, and RNA-Seq), as well as testing for pre-clinical , biomarkers of the pathobiological processes of CVD or CVD phenotypes (e.g. coronary artery calcification, microalbuminuria, leukocyte telomeres, or vascular dysfunction). It is anticipated that these deep sequencing efforts will yield novel ancestry-related DNA variants associated with the CVD phenotypes; yet with unclear biological significance in elucidating racial disparities in CVD. Accordingly, our protocol also includes a Genotype-to-Phenotype (G2P) component that re- contacts subsets of the cohort based on their genotype (e.g. APOL1 chronic kidney disease risk alleles) for a call-back visit for more in-depth phenotyping and characterization of the potential effect of the DNA variant of interest on human systems biology. In some cases family members of the proband may also be invited to participate in these G2P studies to further characterize the biological significance of these putative functional DNA variants of interest.

The primary outcome variables involve well established CVD phenotypes: 1) CVD risk factors (e.g. hypertension, dyslipidemia), 2) markers of pre-clinical CVD (i.e. coronary artery calcification, coronary plaque burden by cardiac CT angiography (CTA), carotid plaque burden by 3D ultrasound, vascular dysfunction, microalbuminuria, C-reactive protein, Vitamin D levels). The protocol will assess exposures associated with CVD and relevant covariates including: 1) social determinants (e.g. socioeconomic status (SES), perceived stress, discrimination, and depression); 2) environmental factors such as neighborhood characteristics (geospatial features of healthy lifestyles [e.g. walkability]) and 3) behavioral factors (e.g. diet, physical activity). The G2P callback visit protocol will involve additional measures of in-depth phenotyping that include: 1) peripheral immune cell phenotyping (e.g. T-cell, monocyte subsets); 2) blood/immune cell RNAseq; 3) iPSC cell line generation (endothelial; vascular smooth muscle cells) and analysis of cardiovascular cell systems biology; 4) HDL proteome analysis, 5) FDG PET/CT and/or PET/MRI scan (vascular inflammation) 6) echocardiography, 7) bisulfite sequencing for identifying sites of DNA methylation, and 8) chromatin immunoprecipitation followed by sequencing (Chip-Seq) for identifying sites of histone modification. It is anticipated that this multi-level, multi-dimensional analysis of genomic and phenotypic characteristics of AA will advance our understanding of the bio-social determinants of the intragroup variance and the increased overall burden of CVD observed among AA.

ELIGIBILITY:
* INCLUSION CRITERIA:

Community-based self-identified (non-institutionalized), US-born, African American men and women age 21-65 will be included in the study. This criterion is inclusive of self-identified AA of both Hispanic and non-Hispanic ethnicity.

EXCLUSION CRITERIA:

Pregnant women are excluded from all aspects of the protocol. Adults who are unable to provide informed consent will be excluded. There are various reasons for excluding pregnant women from all protocol activities. It is well established that many of the primary and secondary study outcome variables and covariates being assessed by the protocol are significantly influenced by the pregnant state. For example pregnancy is known to affect multiple key study variables such as: blood pressure, endothelial function, vascular compliance/stiffness, body mass index, glucose-insulin metabolism and various neurohumoral factors involved in cardiovascular homeostasis. Similarly, pregnancy may have a confounding effect on important behavioral and psycho-social parameters under study (e.g. diet, sleep habits, physical activity, perceived stress, depression). Moreover, it is anticipated that a long-term objective of the study is to "call-back" many GENE-FORECAST participants for either follow-up and/or serial, longitudinal assessments of certain key parameters. It is therefore essential that the initial baseline evaluation not involve a transient condition such as pregnancy that has such profound effects on the cardio-metabolic phenotype under study. Neonates are excluded because they are less than the age of 21 years.

Non-English speaking African Americans and those not born in the United States will be excluded. These individuals will be excluded because the exposure to social determinants experienced by African Americans born in the US differs from that of Africans born elsewhere and because the survey instruments in this protocol have only been verified in English speaking African-Americans. Furthermore, African immigrants are likely to have metabolic and cardiovascular profiles that are distinct from African Americans, and this could be a source of uncharacterized confounding factors. Those with severe and disabling co-morbidities associated with end-stage CVD will be excluded such as a recent history of hospitalization for manifestations of cardiovascular disease. More specifically, patients with a history of stroke, heart attack and/or heart failure in the past 12 months will be excluded. Nursing females will be excluded from FGD PET/CT and/or PET/MRI. Participants with pacemakers and/or any history of metal device implantation and/or metal in their body will be excluded from MRI according to clinical center guidelines. Participants with implanted electronic medical device will be excluded from percent body fat measurement. For CTA, patients with known allergic reaction to contrast will not be given contrast. Diabetic patients taking metformin will be excluded from receiving CTA IV contrast agents. Patients with renal failure (eGFR<60) will not be given either MRI or CTA IV contrast. Adults who are or may be unable to consent are excluded due to their lack of knowledge to study components.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary Clinical and community sample
Sampling Method: Non-Probability Sample
Enrollment: 670 (Actual)
Dates: Start 2014-07-23 (Actual); Primary Completion 2024-03-08 (Actual); Study Completion 2024-03-08 (Actual)

PRIMARY OUTCOMES:
Our objective is to develop a community-based cohort and novel genomic science resource for defining the biological significance of ancestry-related genomic variation in African-Americans within the GENE-FORECAST(R): GENomics, Environmental Fact... | one time assessment
  Our objective is to develop a community-based cohort and novel genomic science resource for defining the biological significance of ancestry-related genomic variation in African-Americans within the GENE-FORECAST(R): GENomics, Environmental FactORs and the Social DEterminants of Cardiovascular Disease in African Americans Study.

CONTACTS AND LOCATIONS:
Overall Officials: Tiffany M Powell-Wiley, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (2):
- United States (2):
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - Southern Research Group, Jackson, Mississippi

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2014-HG-0048.html